CLINICAL TRIAL: NCT04571710
Title: A Phase 2 Study of Pyrotinib in Patients With Advanced/ Metastatic HER2-Altered Biliary Tract Cancers Who Have Failed One or Two Prior Lines of Therapies
Brief Title: A Trial of SHR1258 in Patients With Biliary Tract Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor's R&D strategy is adjusted.
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-BLTN-II-BTC
Record Dates: First submitted 2020-09-17; First posted 2020-10-01 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Intervention: Drug: SHR1258 400mg
  Interventions: Drug: SHR1258

INTERVENTIONS:
Drug: SHR1258 — Drug: SHR1258 400mg

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR1258 in subjects with advanced/ metastatic HER2-altered biliary tract cancers

ELIGIBILITY:
Inclusion Criteria:

* enrollment into the study:

  1. Signed and dated written informed consent which is approved by Institutional Review Board (IRB)/Ethics Committee (EC), willing and able to comply with scheduled treatment, all examinations at study visits, and other study procedures.
  2. Male or female, ≥18 years old.
  3. Histologically or cytologically confirmed (at a local laboratory) BTC
  4. Received up to two prior regimen of systemic therapy for advanced disease, including 1 gemcitabine-containing regimen, and experienced disease progression after or developed intolerance to the most recent prior therapy.
  5. Sufficient tumor tissue samples (archival or fresh biopsy samples) will be provided by all subjects prior to the administration of pyrotinib (for retrospective confirmation of HER2 alteration through a central laboratory if applicable).
  6. Must have measureable disease per RECIST v1.1. The definition of CT or MRI measurable lesion as the target lesion: according to RECIST v1.1, the long diameter of such lesion should be ≥ 10 mm by the CT scan or the short diameter of enlarged lymph nodes ≥ 15 mm.
  7. The laboratory test values must meet the functional level of important organs/systems meets
  8. ECOG-PS (see Appendix 2): 0 - 1.
  9. If subjects have active hepatitis B virus (HBV) infection: HBV- deoxyribonucleic acid (DNA) must be < 500 IU/mL and are willing to receive antiviral therapy throughout the study; subjects with positive hepatitis C (HCV) ribonucleic acid (RNA) must receive antiviral therapy in accordance with the local standard treatment guideline and have ≤ CTCAE Grade 1 elevated hepatic function.
  10. Women of childbearing potential (WOCBP) must have a serum pregnancy test within 7 days before the first dose and the result is negative. WOCBP and male subjects whose partners are WOCBP must agree to use effective contraception method during the study period and within 8 weeks after the last dose of study medication.

Exclusion Criteria:

* Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Signed and dated written informed consent which is approved by Institutional Review Board (IRB)/Ethics Committee (EC), willing and able to comply with scheduled treatment, all examinations at study visits, and other study procedures.
2. Male or female, ≥18 years old.
3. Histologically or cytologically confirmed (at a local laboratory) BTC
4. Received up to two prior regimen of systemic therapy for advanced disease, including 1 gemcitabine-containing regimen, and experienced disease progression after or developed intolerance to the most recent prior therapy.
5. Sufficient tumor tissue samples (archival or fresh biopsy samples) will be provided by all subjects prior to the administration of pyrotinib (for retrospective confirmation of HER2 alteration through a central laboratory if applicable).
6. Must have measureable disease per RECIST v1.1. The definition of CT or MRI measurable lesion as the target lesion: according to RECIST v1.1, the long diameter of such lesion should be ≥ 10 mm by the CT scan or the short diameter of enlarged lymph nodes ≥ 15 mm.
7. The laboratory test values must meet the functional level of important organs/systems meets
8. ECOG-PS (see Appendix 2): 0 - 1.
9. If subjects have active hepatitis B virus (HBV) infection: HBV- deoxyribonucleic acid (DNA) must be < 500 IU/mL and are willing to receive antiviral therapy throughout the study; subjects with positive hepatitis C (HCV) ribonucleic acid (RNA) must receive antiviral therapy in accordance with the local standard treatment guideline and have ≤ CTCAE Grade 1 elevated hepatic function.
10. Women of childbearing potential (WOCBP) must have a serum pregnancy test within 7 days before the first dose and the result is negative. WOCBP and male subjects whose partners are WOCBP must agree to use effective contraception method during the study period and within 8 weeks after the last dose of study medication.

Exclusion Criteria:

Subjects presenting with any of the following will not be enrolled into the study:

1. Prior receipt of HER2-targeted therapy.
2. Concurrent anticancer therapy, other than the therapies being tested in this study.
3. Radiation therapy administered within 2 weeks of first dose of study treatment.
4. Laboratory values at screening outside the protocol-defined range.
5. Clinically significant or uncontrolled cardiac disease.
6. Target disease exclusion criteria:

1) Malignant tumors with other pathological types, such as mixed cancer, double primary cancers.

2) Medical history of other active malignancies within last 5 years. 3) Subjects with active central nervous system (CNS) metastases are excluded. Subjects with history or evidence of current leptomeningeal metastases are excluded.

4) By the date of first dose of study treatment, the washout period of previous drug treatment / medical intervention does not meet the following requirements 7. Medical history exclusion criteria:

1. Severe cardiac disease
2. Prior to the first dose of study treatment, patients with the following conditions: inability to swallow, chronic diarrhea, intestinal obstruction, gastrointestinal perforation or gastrectomy, colitis or other diseases or special conditions that affect drug administration and absorption.
3. Prior to the first dose of study treatment, patients with severe effusions with clinical symptoms
4. Symptoms of severe infection or evidence for microbiological/viral diagnosis.
5. Congenital or acquired immunodeficiency (e.g., human immunodeficiency virus [HIV] infection).

8. History of allergy to the study drugs or components. 9. Pregnancy or breastfeeding. 10. Concomitant treatments exclusion criteria:

1. Within 2 weeks prior to the first dose of study treatment, or during the study period, patients receive or are anticipated to receive continuous strong CYP3A4 inducers or inhibitors, P-gp inhibitors.

11. Others:

1. Per investigator's judgment, other diseases or laboratory evidence that would cause serious threats to the safety of the patients, or which are not in the best interest of the patient to participate in the study are excluded
2. Per investigator's judgment, other situations that may confuse the study results or would affect the subjects' ability to comply with study procedures are excluded, such as alcoholism, drug abuse, criminal detention, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Objective response rate | up to 2 years
  Objective response rate (ORR) evaluated by Blinded Independent Radiology Review Committee (BIRC) based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
DOR | up to 2 years
  Duration of response
DCR | up to 2 years
  Disease Control Rate
PFS | up to 2 years
  Progression-Free-Survival
OS | up to 2 years
  overall survival
AEs+SAEs | from the first drug administration to within 28 days for the last SHR1258 dose
  Adverse event
Cmax | up to 2 years
  Peak Plasma Concentration